CLINICAL TRIAL: NCT04911699
Title: Trajectory Analysis of Symptom Distress and Cancer-related Fatigue After Adjuvant Chemotherapy in Breast Cancer Female: an Prospective Study
Brief Title: Trajectory Analysis of Symptom Distress and Cancer-related Fatigue After Adjuvant Chemotherapy in Breast Cancer Female
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Tsai-Wei Huang, School of Nursing, Taipei Medical University
Other Study IDs: symptom of breast cancer
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Symptom Distress During Breast Cancer Treatment
Keywords: Breast cancer; cancer related fatigue; symptom distress; insomnia; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- breast adenocarcinoma: 1. The surgical pathological tissue report confirms the diagnosis of breast adenocarcinoma women with stage I~III
  2. Those who are admitted to the hospital and receive adjuvant chemotherapy for the first time.
  3. Age (inclusive) over 20 years old.
  Interventions: Behavioral: breast adenocarcinoma receiving chemotherapy
- Control: 1. The surgical pathological tissue report establishes women diagnosed as stage 0 to stage III breast cancer
  2. Those who are admitted to the hospital to receive anti-hormonal drug treatment.
  3. Age (inclusive) over 20 years old.
  Interventions: Behavioral: Control-for

INTERVENTIONS:
Behavioral: breast adenocarcinoma receiving chemotherapy — for chemotherapy
  Groups: breast adenocarcinoma
Behavioral: Control-for — hormonal drug treatment
  Other Names: hormonal drug treatment
  Groups: Control

SUMMARY:
When receiving adjuvant chemotherapy, a variety of symptoms will appear and it is very painful. These symptoms occur at the same time and are related to each other. The symptom distress may affect the patient's compliance with adjuvant chemotherapy and whether the adjuvant chemotherapy can be completed on schedule. Among the symptoms of trouble, cancer-related fatigue is the most common, and the incidence can be as high as 99%. In this study, I want to track the population of breast cancer patients receiving adjuvant chemotherapy, and women in the control group who receive only anti-hormonal breast cancer or carcinoma in situ. During the treatment period, at different time points, it also collects subjective symptom distress changes and changes. The study aimed cancer-related exhaustion is measured to gain a deeper understanding of the effects of symptom troubles suffered by patients during treatment. We also hoped that in the future, it can be provided to colleagues in clinical work and can be given to breast cancer patients receiving adjuvant chemotherapy and increased holistic care quality.

ELIGIBILITY:
Inclusion Criteria:

1. The surgical pathological tissue report confirms that the diagnosis is zero stage breast carcinoma in situ women and stage I~III Breast cancer women.
2. Those who are admitted to the hospital for the first time adjuvant chemotherapy or hormonal therapy.
3. Age (inclusive) over 20 years old

Exclusion Criteria:

1. Women with breast cancer who are unconscious or unable to express.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast carcinoma in situ women and stage I~III Breast cancer women receiving therapy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-29 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Trajectory of Symptom distress | T0 to T6, T0 pre chemotherapy; T1, chemotherapy 1 month; T2, chemotherapy 2 month; T3, chemotherapy 3 month;T4, chemotherapy 4 month;T5, chemotherapy 5 month;T6, chemotherapy 6 month;
  Edmonton Symptom Assessment Scale, ESAS; including nine symptoms, one symptom range from 0-10, total score 0-90.
Trajectory of fatigue | T0 to T6, T0 pre chemotherapy; T1, chemotherapy 1 month; T2, chemotherapy 2 month; T3, chemotherapy 3 month;T4, chemotherapy 4 month;T5, chemotherapy 5 month;T6, chemotherapy 6 month;
  Brife fatigue inventory, BFI; including nine items, total score 0-10.
Trajectory of distress temperature | T0 to T6, T0 pre chemotherapy; T1, chemotherapy 1 month; T2, chemotherapy 2 month; T3, chemotherapy 3 month;T4, chemotherapy 4 month;T5, chemotherapy 5 month;T6, chemotherapy 6 month;
  Distress Thermometer, DT; range from 0-10.
Trajectory of Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | T0 to T6, T0 pre chemotherapy; T1, chemotherapy 1 month; T2, chemotherapy 2 month; T3, chemotherapy 3 month;T4, chemotherapy 4 month;T5, chemotherapy 5 month;T6, chemotherapy 6 month;
  FACT-B;multidimensional questionnaire with 37 items that build 5 dimensions (subscales) when using a 5-point Likert scale. (from 0, not at all through 4, very much) that constitute 5 dimensions.
Trajectory of PHQ-4: Validated Screening Tool for Anxiety and Depression | T0 to T6, T0 pre chemotherapy; T1, chemotherapy 1 month; T2, chemotherapy 2 month; T3, chemotherapy 3 month;T4, chemotherapy 4 month;T5, chemotherapy 5 month;T6, chemotherapy 6 month;
  PHQ-4;PHQ-4 Scoring: Total score ranges from 0 to 12, with categories of psychological distress as follows:
  None: 0-2; Mild: 3-5; Moderate: 6-8; Severe: 9-12; Anxiety subscale = sum of items 1 and 2 (score range: 0 to 6) Depression subscale = sum of items 3 and 4 (score range: 0 to 6) On each subscale, a score of 3 or greater is considered positive for screening purposes.
Trajectory of ISI: Insomnia Severity Index | T0 to T6, T0 pre chemotherapy; T1, chemotherapy 1 month; T2, chemotherapy 2 month; T3, chemotherapy 3 month;T4, chemotherapy 4 month;T5, chemotherapy 5 month;T6, chemotherapy 6 month;
  (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia. ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia.11,24 The usual recall period is the "last month" and the dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).